CLINICAL TRIAL: NCT01146587
Title: Robot Assisted Therapy for Acute Stroke Patients: a Comparative Study of GangTrainer GT I, Lokomat System and Conventional Physiotherapy
Brief Title: Comparative Study of GangTrainer GT1, Lokomat and Conventional Physiotherapy
Acronym: galop
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: GangTrainer GT1 is not state of the art anymore for the principal Invesigator
Sponsor: Research Department for Neurorehabilitation South Tyrol (Other)
Collaborators: Privatklinik Villa Melitta (Other); Hochzirl Hospital (Other); Krankenhaus Bozen (Other); Krankenhaus Brixen (Other); Krankenhaus Meran (Other); Krankenhaus Bruneck (Other); Claudiana Landesfachhochschule (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GT-LK-PT
Record Dates: First submitted 2010-06-14; First posted 2010-06-17 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Stroke, Acute
Keywords: Stroke; Robotics; Gait; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- GangTrainer GT1 (Experimental): First supratentorial non ambulatory stroke patients (ischaemic, haemorrhagic or ICH) with a hemiparesis and stroke onset from 3 - 12 weeks undergo robotic treatment with the Gangtrainer GT1 for 30 minutes of gross therapy time every workday for a 8 weeks period
  Interventions: Device: GangTrainer GT1
- Lokomat (Experimental): First supratentorial non ambulatory stroke patients (ischaemic, haemorrhagic or ICH) with a hemiparesis and stroke onset from 3 - 12 weeks undergo robotic treatment with the Lokomat for 30 minutes of gross therapy time every workday for a 8 weeks period
  Interventions: Device: Lokomat
- Conventional Physiotherapy (Active Comparator): First supratentorial non ambulatory stroke patients (ischaemic, haemorrhagic or ICH) with a hemiparesis and stroke onset from 3 - 12 weeks undergo a conventional physiokinetherapeutic treatment session for 30 minutes of gross therapy time every workday for a 8 weeks period
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Device: GangTrainer GT1 — 30 minutes of treatment on the GangTrainer GT1 and 30 minutes of Conventional Physiotherapy every workday for 8 weeks
  Other Names: Group A
  Arms: GangTrainer GT1
Device: Lokomat — 30 minutes of treatment on the Lokomat and 30 minutes of Conventional Physiotherapy every workday for 8 weeks
  Other Names: Group B
  Arms: Lokomat
Other: Conventional Physiotherapy — 60 minutes of Conventional Physiotherapy every workday for 8 weeks
  Other Names: Group C
  Arms: Conventional Physiotherapy

SUMMARY:
The GangTrainer GT I and the Lokomat have proven their effectiveness on stroke Patients, but a comparison on the same controlled study population has not been made so far. Aim of the study will not only be to establish which device will work better on acute, non ambulatory stroke Patients in terms of regain of gait ability and motor function, but also clinical matters, like the efficacy of the treatment period. As a result of the trial it should be highlighted which kind of therapy has to be suggested for Patients comparable to the study population. A significant better outcome of one device in regard to the other will suggest to use one device more than the other for future treatments.

DETAILED DESCRIPTION:
A total of 120 Patients will be enroled in the study and divided into 2 treatment and 1 control group. Enroled Patients will all be first supratentorial non ambulatory stroke patients (ischaemic, haemorrhagic or ICH) with a hemiparesis and stroke onset from 3 - 12 weeks.

Theywill undergo either robotic treatment with the Gangtrainer GT1 or the Lokomat in one of the 2 treatment groups for 30 minutes of gross therapy time every workday for a 8 weeks period if they are in the treatment group, or conventional physiokinetherapy for 30 minutes of gross therapy time every workday for a 8 weeks period if they are in the control group.

Primary outcome will be the Functional Ambulation Category (FAC) assessed at enrolment, after 4 weeks after 8 weeks and at 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* First supratentorial stroke (ischaemic, haemorrhagic or ICH) resulting in a hemiparesis
* Interval from stroke 3 - 12 weeks
* Non ambulatory (FAC < 3)
* Free sitting on bedside for 1 minute, both feet on the floor, ev. holding on bedside by hands
* Barthel Index 25 - 65

Exclusion Criteria:

* Unstable cardiovascular system (in case of doubt, only after approval by a internist)
* Manifested heart diseases like labile compensated cardiac insufficiency (NYHA III), angina pectoris, myocardial infarction 120 days before study onset, cardiomyopathy, severe cardiac arrhythmia
* Severe joint misalignment (severe constriction of movement for hip, knee and/or ankle: more than 20° fixed hip and knee extension deficit, or more than 20° fixed plantar flexion of the ankle
* Severe cognitive dysfunction, which does not allow for comprehension of the aims of this study
* Severe neurological or orthopaedic diseases (like polio, Parkinson´s disease), which massively affect the mobility
* Deep vein thrombosis
* Severe osteoporosis
* Malignant tumour diseases

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulation Category (FAC) | after 8 weeks

SECONDARY OUTCOMES:
Barthel Index (BI) | at week 1
Barthel Index (BI) | after 4 weeks
Barthel Index (BI) | after 8 weeks
Barthel Index (BI) | after 24 weeks
Rivermead Mobility Index (RMI) | at week 1
Rivermead Mobility Index (RMI) | after 4 weeks
Rivermead Mobility Index (RMI) | after 8 weeks
Rivermead Mobility Index (RMI) | after 24 weeks
10 metres Walking Test | at week 1
10 metres Walking Test | after 4 weeks
10 metres Walking Test | after 8 weeks
10 metres Walking Test | after 24 weeks
6 Minutes Walking Test on the Floor | at week 1
6 Minutes Walking Test on the Floor | after 4 weeks
6 Minutes Walking Test on the Floor | after 8 weeks
6 Minutes Walking Test on the Floor | after 24 weeks
6 Minutes Walking Test on the Treadmill with Body Weight Support | at week 1
6 Minutes Walking Test on the Treadmill with Body Weight Support | after 4 weeks
6 Minutes Walking Test on the Treadmill with Body Weight Support | after 8 weeks
6 Minutes Walking Test on the Treadmill with Body Weight Support | after 24 weeks
Medical Research Council (MRC) | at week 1
Medical Research Council (MRC) | after 4 weeks
Medical Research Council (MRC) | after 8 weeks
Medical Research Council (MRC) | after 24 weeks
Modified Ashworth Scale (mAS) | at week 1
Modified Ashworth Scale (mAS) | after 4 weeks
Modified Ashworth Scale (mAS) | after 8 weeks
Modified Ashworth Scale (mAS) | after 24 weeks
Rivermead Visual Gait Assessment (RVGA) | at week 1
Rivermead Visual Gait Assessment (RVGA) | after 8 weeks
Rivermead Visual Gait Assessment (RVGA) | after 24 weeks
EuroQol 5 Dimensions (EQ-5D) | at week 1
EuroQol 5 Dimensions (EQ-5D) | after 8 weeks
EuroQol 5 Dimensions (EQ-5D) | after 24 weeks
modified emory Functional Ambulation Profile (meFAP) | at week 1
modified emory Functional Ambulation Profile (meFAP) | after 4 weeks
modified emory Functional Ambulation Profile (meFAP) | after 8 weeks
modified emory Functional Ambulation Profile (meFAP) | after 24 weeks
Functional Ambulation Category (FAC) | at week 1
Functional Ambulation Category (FAC) | after 4 weeks
Functional Ambulation Category (FAC) | after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Waldner, MD, Principal Investigator — Privatklinik Villa Melitta; Christopher Tomelleri, MSc, Study Chair — Privatklinik Villa Melitta; Leopold Saltuari, MD PhD, Study Director — Hochzirl Hospital
Locations (7):
- Hochzirl Hospital, Hochzirl, Tyrol, Austria
- Italy (6):
  - Claudiana Landesfachhochschule, Bolzano, Südtirol
  - Krankenhaus Bozen, Bolzano, Südtirol
  - Privatklinik Villa Melitta, Bolzano, Südtirol
  - Krankenhaus Brixen, Brixen, Südtirol
  - Krankenhaus Bruneck, Bruneck, Südtirol
  - Krankenhaus Meran, Meran, Südtirol

REFERENCES:
- [Background] Kolominsky-Rabas PL, Heuschmann PU. [Incidence, etiology and long-term prognosis of stroke]. Fortschr Neurol Psychiatr. 2002 Dec;70(12):657-62. doi: 10.1055/s-2002-35857. German. PMID 12459947
- [Background] Barbeau H, Visintin M. Optimal outcomes obtained with body-weight support combined with treadmill training in stroke subjects. Arch Phys Med Rehabil. 2003 Oct;84(10):1458-65. doi: 10.1016/s0003-9993(03)00361-7. PMID 14586912
- [Background] Hidler J, Nichols D, Pelliccio M, Brady K, Campbell DD, Kahn JH, Hornby TG. Multicenter randomized clinical trial evaluating the effectiveness of the Lokomat in subacute stroke. Neurorehabil Neural Repair. 2009 Jan;23(1):5-13. doi: 10.1177/1545968308326632. PMID 19109447
- [Background] Pohl M, Werner C, Holzgraefe M, Kroczek G, Mehrholz J, Wingendorf I, Hoolig G, Koch R, Hesse S. Repetitive locomotor training and physiotherapy improve walking and basic activities of daily living after stroke: a single-blind, randomized multicentre trial (DEutsche GAngtrainerStudie, DEGAS). Clin Rehabil. 2007 Jan;21(1):17-27. doi: 10.1177/0269215506071281. PMID 17213237
- [Background] Regnaux JP, Saremi K, Marehbian J, Bussel B, Dobkin BH. An accelerometry-based comparison of 2 robotic assistive devices for treadmill training of gait. Neurorehabil Neural Repair. 2008 Jul-Aug;22(4):348-54. doi: 10.1177/1545968307310050. Epub 2007 Dec 11. PMID 18073325
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Baer HR, Wolf SL. Modified emory functional ambulation profile: an outcome measure for the rehabilitation of poststroke gait dysfunction. Stroke. 2001 Apr;32(4):973-9. doi: 10.1161/01.str.32.4.973. PMID 11283399
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Collen FM, Wade DT, Robb GF, Bradshaw CM. The Rivermead Mobility Index: a further development of the Rivermead Motor Assessment. Int Disabil Stud. 1991 Apr-Jun;13(2):50-4. doi: 10.3109/03790799109166684. PMID 1836787
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Lord SE, Halligan PW, Wade DT. Visual gait analysis: the development of a clinical assessment and scale. Clin Rehabil. 1998 Apr;12(2):107-19. doi: 10.1191/026921598666182531. PMID 9619652
- See also: Participating Centre for the interventions GangTrainer GT1 and Conventional Physiotherapy — http://www.villamelitta.it
- See also: Participating Centre for the interventions Lokomat and Conventional Physiotherapy — http://neuro-hochzirl.tilak.at
- See also: Participating Centre responsible for the blinded rating of the visual gait analysis — http://www.claudiana.bz.it/